CLINICAL TRIAL: NCT06939842
Title: The Effect of Menthol Ice and Frozen Saline Applications on Patients' Thirst and Sore Throat After Lumbar Disc Surgery
Brief Title: The Effect of Menthol Ice and Frozen Saline Applications After Lumbar Disc Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kübra TUNCEL, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IUC-SN-KT-01
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-04

CONDITIONS: Thirst; Sore Throat
Keywords: Lumbar Disc Disease; Thirst; Menthol; Ice
MeSH Terms: conditions — Pharyngitis; Intervertebral disc disease

STUDY DESIGN:
Intervention Model Description: Three groups with control group (The study was planned as an open-label, randomized, controlled, parallel group interventional study. Participants will be randomly assigned to groups.)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Menthol ice group (Experimental): The menthol ice group will be given menthol ice by the researcher.
  Interventions: Other: Menthol ice
- Frozen saline group (Experimental): The frozen saline group will be given frozen saline by the researcher.
  Interventions: Other: Frozen saline
- Control group (Other): There will be no intervention to the control group. Routine practices of the clinic (moisturizing the lips with wetgauze, cotton or tissue) will be performed by the nurses of the Surgery Clinics.
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: Menthol ice — When patients are brought from the operating theatre to the surgical clinic, patients will be waited until they are able to communicate. In the first stage, after filling in the Patient Identification Form before the intervention, thirst status with Perioperative Thirst Discomfort Scale (PTDS) and sore throat status with the Numerical Pain Scale (NPS) will be evaluated. In the second stage, evaluation will be made according to the Safety Protocol for the Management of Immediate Postoperative Thirst and menthol ice will be applied if the patients meet the criteria in the protocol. Thirst will be re-evaluated with PTDS and sore throat will be re-evaluated with NPS at 30th and 60th minutes after the first application. Immediately after this evaluation, menthol ice will be applied for the second time. After the second application, thirst will be re-evaluated with PTDS at 30th and 60th minutes and sore throat will be re-evaluated with NPS.
  Arms: Menthol ice group
Other: Frozen saline — When patients are brought from the operating theatre to the surgical clinic, patients will be waited until they are able to communicate. In the first stage, after filling in the Patient Identification Form before the intervention, thirst status with Perioperative Thirst Discomfort Scale (PTDS) and sore throat status with the Numerical Pain Scale (NPS) will be evaluated. In the second stage, evaluation will be made according to the Safety Protocol for the Management of Immediate Postoperative Thirst and frozen saline will be applied if the patients meet the criteria in the protocol. Thirst will be re-evaluated with PTDS and sore throat will be re-evaluated with NPS at 30th and 60th minutes after the first application. Immediately after this evaluation, frozen saline will be applied for the second time. After the second application, thirst will be re-evaluated with PTDS at 30th and 60th minutes and sore throat will be re-evaluated with NPS.
  Arms: Frozen saline group
Other: No Interventions — When patients are brought from the operating theatre to the surgical clinic, patients will be waited until they are able to communicate. In the first stage, after filling in the Patient Introduction Form before the intervention, thirst status with Perioperative Thirst Discomfort Scale (PTDS) and sore throat status with Numerical Pain Scale(NPS) will be evaluated. Patients in the control group will be waited for approximately 10 minutes, taking into account the application times in the intervention groups. No intervention will be applied during the waiting period. After 10 minutes of waiting time, thirst will be re-evaluated with PTDS and sore throat will be re-evaluated with NPS at 30th and 60th minutes. Considering the 2nd application time in the intervention groups, it will be waited again for approximately 10 minutes without any intervention. After the waiting period, thirst will be re-evaluated with PTDS at 30th and 60th minutes and sore throat will be re-evaluated with NPS.
  Arms: Control group

SUMMARY:
The aim of the study was to determine the effect of postoperative menthol ice and frozen saline applications on thirst and sore throat in patients undergoing lumbar disc surgery.

DETAILED DESCRIPTION:
In the postoperative period, patients become susceptible to many complications that may develop due to general anaesthesia, endotracheal intubation, surgical intervention and clinical conditions. One of the conditions that patients experience quite intensely in the postoperative period and which is usually ignored in clinics is the feeling of thirst. Another problem that may occur in patients undergoing surgery under general anaesthesia is discomfort due to endotracheal intubation. Patients may experience problems such as sore throat, hoarseness, difficulty swallowing and dry throat in the postoperative period due to endotracheal intubation. Diagnosis and control of postoperative thirst and sore throat contribute to patient comfort and prevention of complications. This study is considered important because it draws attention to postoperative thirst and sore throat, a problem that surgical patients have.

ELIGIBILITY:
Inclusion Criteria:

* Knowing how to read, write and speak Turkish
* Having no obstacle in understanding and communicating the information given
* Agreeing to participate in the research verbally and in writing after being informed about the research
* Ages 18 and over
* Those who underwent surgery under general anesthesia
* Those who have not yet started oral intake in the postoperative period
* Without menthol allergy
* According to the American Society of Anesthesiologists (ASA) classification; Class I, II and III, Normal healthy patient (ASA I); Patient with mild systemic disease (ASA II); Patient with serious systemic disease that does not affect daily activities (ASA III)
* Having no sore throat before surgery
* As a result of the evaluation made with the Safety Protocol for Management Thirst in the Early Postoperative Period , patients who provide appropriate conditions for ice application (the individual must be conscious and oriented after the surgery, the airway must be open with coughing, swallowing and breathing, and there is no nausea or vomiting)

Exclusion Criteria:

* Those who have severe nausea and vomiting at the time of application
* Those with a change in consciousness status/acute confusion after surgical intervention
* Those with chronic disease/diseases related to Ear-Nose-Throat Diseases
* Patients with difficult intubate
* Patients with psychiatric problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Total Score on the Perioperative Thirst Discomfort Scale | Baseline (pre-intervention), and at 30 and 60 minutes after each of two interventions (total of 5 time points within 2 hours post-op).
  The Perioperative Thirst Discomfort Scale is a 6-item self-report instrument. It uses a 3-point Likert response format with each item rated as: 0 = Did not disturb, 1 = Somewhat disturbed, and 2 = Very disturbed. The total score ranges from 0 to 12, with higher scores indicating greater perioperative thirst discomfort. The scale has no sub-dimensions. It is used to quantitatively assess patients' perceived thirst discomfort during the perioperative period.

SECONDARY OUTCOMES:
Throat Pain Intensity as Measured by the Numerical Pain Scale | Baseline (pre-intervention), and at 30 and 60 minutes after each of two interventions (total of 5 time points within 2 hours post-op).
  Throat pain intensity was assessed using a Numerical Pain Scale ranging from 0 to 10, where 0 indicates no throat pain and 10 indicates the worst throat pain imaginable. Participants rated their throat pain by selecting a number that best described its intensity at the time of assessment. The Numerical Pain Scale is a validated and widely used tool for measuring subjective pain.
Eligibility for Oral Hydration Administration According to the Safety Protocol for Management Thirst in the Immediate Postoperative Period | Baseline (pre-intervention) (total of one time point within post-op period)
  The Safety Protocol for Thirst Management in the Immediate Postoperative Period is a checklist-based protocol designed to evaluate whether patients in the early post-anesthesia period are eligible for oral water or ice administration. The protocol assesses key clinical criteria such as level of consciousness, airway patency, and presence of nausea or vomiting. Only patients who meet all the checklist criteria are considered suitable for oral water or ice administration.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra TUNCEL, PhD-candidate, Principal Investigator — Istanbul University-Cerrahpasa Institute of Graduate Studies
Locations (1):
- Istanbul University-Cerrahpasa Institute of Graduate Studies, Istanbul, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No